CLINICAL TRIAL: NCT04923217
Title: Assessing Quality of Life and Sexual Function in Vaginal Aplasia Patients After Neovaginal Surgical Procedure by Davydov Method
Brief Title: Quality of Life and Sexual Function in Vaginal Aplasia Patients After Davydov Procedure
Status: Completed | Type: Observational
Sponsor: School of Medicine - Vietnam National University at Ho Chi Minh city (Other)
Collaborators: Tu Du Hospital (Other Government); University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thanh Le Trung Quoc, Principle investigator, School of Medicine - Vietnam National University at Ho Chi Minh city
Other Study IDs: 50/HĐĐĐ-ĐHYD
Record Dates: First submitted 2021-05-21; First posted 2021-06-11 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome; Quality of Life; Sexual Function Disturbances
MeSH Terms: conditions — Mullerian aplasia; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mayer-Rokitansky-Kuster-Hauser(MRKH) syndrome is described as absence or underdevelopment of vagina and uterus. This condition is extremely rare congenital malformation that affects one in every 5000 female births. Medical management of MRKH syndrome includes the creation of a neovagina using nonsurgical or surgical procedure. In Vietnam, since 2014, Davydov technique has been used to create neovagina for patients with MRKH syndrome at Tu Du hospital which is the biggest obstetric and gynecological hospital in south of Vietnam. However, the effectiveness of this surgical approach on patient's life and sexual activity hasn't been assessed. The objective of this study is to assess the quality of life, the psychological impact and the sexual function of Vietnamese women with MRKH syndrome after Davydov surgical procedure.

DETAILED DESCRIPTION:
This study will be conducted at Tu Du Hospital, Ho Chi Minh City, Vietnam. Female patients diagnosed with Mayer-Rokitansky-Kuster-Hauser (MRKH) syndrome were performed the Davydov procedure to create neovagina at the Anaesthesia and Intensive care department, Tu Du hospital. Based on the Department of Anaesthesia and Intensive care data, a list of potentially eligible patients who underwent Davydov surgery at least six months was made. Because of the impact of the Covid 19 pandemic, the patients could not come to the hospital, so the research team decided to interview the participants online. According to this list, patients will be contacted by telephone to set up an online appointment to assess the effectiveness of the Davydov procedure. The informed consent will be sent by email or mail to the patients who accepted to participate in our research before the enrolment. On appointment day, the investigator will make group telecommunication by an application on cell phone or computer. Efficacy of Davydov procedure according to the functional aspect: the psychological doctors assess the impact of patient's neovagina on life and sexual function through questionnaires involving World Health Organization Quality of life Scale (WHOQoL-BREF), Female Sexual Function Index (FSFI) and self-composed qualitative questionnaire. The interview with a patient will be held individually and conducted by the psychological doctor. The participants will be requested to record the conversation. Because MRKH syndrome is a rare condition, the investigators take all patients who are suitable to inclusion criteria and accept participating in our research.

ELIGIBILITY:
Inclusion Criteria:

* Aged equal or more than 18.
* Diagnosed vaginal agenesis and underwent Davydov procedure to create neovagina at least 6 months.
* Able to listen, understand and answer questions.

Exclusion Criteria:

* Disagreed to participate the research.
* Having any conditions that make patient unable to listen, understand and answer questions.
* Having psychological disturbance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample is patients who underwent Davydov procedure to create neovagina at Tu Du hospital, Ho Chi Minh city, Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life of women with vaginal agenesis after Davydov procedure | From six months after surgery up to the initiation of the study, assessed up to 1 month
  The psychological doctor uses the questionnaire named World Health Organization Quality of Life Scale(WHOQoL-BREF) in the interview to ask patient. The patient's Quality of Life will be assessed based on the WHOQoL-BREF questionnaire 's score. All the results will be collected and calculated subsequently. The raw scores are converted to transformation scores. The first transformation converts scores to range of 4-20 and the second transformation converts domain scores to 0-100 scale. Higher scores reflect better Quality of Life.
Sexual Function of women with vaginal agenesis after Davydov procedure | From six months after surgery up to the initiation of the study, assessed up to 1 month
  The psychological doctor uses the questionnaire named Female Sexual Function Index Scale (FSFI) in the interview to ask patient. The patient's sexual function will be assessed based on the FSFI questionnaire 's score. All the results will be collected and calculated subsequently. The FSFI's minimum total score is 2 and the FSFI's maximum total score is 36. The patient is diagnosed to have sexual dysfunction when the FSFI's total score is less than 26,55.

CONTACTS AND LOCATIONS:
Overall Officials: Lan TN Vuong, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Tu Du Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No